CLINICAL TRIAL: NCT02430363
Title: Phase IIb Trial Evaluations Of The Effectiveness Of Treatment Glioblastoma / Gliosarcoma Through The Suppression Of The PI3K/Akt Pathway In Compared With MK-3475 (Pembrolizumab)
Brief Title: Evaluation Of The Treatment Effectiveness Of Glioblastoma / Gliosarcoma Through The Suppression Of The PI3K/Akt Pathway In Compared With MK-3475
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Medical Research Council (Other Government)
Collaborators: Aarhus University Hospital (Other); NCRI Clinical Studies Groups (Unknown); ECCO - the European CanCer Organisation (Unknown); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ms. Jann Lee, PhD, Medical Research Council
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETIK-W/33-15
Record Dates: First submitted 2015-04-23; First posted 2015-04-30 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Glioblastoma
Keywords: pembrolizumab; MK-3475; Glioblastoma; Gliosarcoma; Suppressor of the PI3K/Akt pathways; Pictilisib; GDC-0941; BEZ235; NVP-BEZ235; Ipatasertib; GDC-0068
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — pembrolizumab; 2-(1H-indazol-4-yl)-6-(4-methanesulfonylpiperazin-1-ylmethyl)-4-morpholin-4-ylthieno(3,2-d)pyrimidine; dactolisib; ipatasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-3475 (Active Comparator): Pembrolizumab (MK-3475) is a humanized monoclonal antibody. Information from these studies suggests that Pembrolizumab (MK-3475) may be beneficial in Glioblastoma / Gliosarcoma.
  * Patients enrolling in phase 1 receive MK-3475 every 3 weeks, with the dose to be determined.
  * MK-3475 will be given intravenously over the course of 30 minutes
  Interventions: Drug: MK - 3475
- Suppressor of the PI3K/Akt pathways (Experimental): Pictilisib (GDC-0941) is a potent inhibitor of PI3Kα/δ. Patients will take the Pictilisib (capsules) orally with food. The dose should be taken every 3 weeks.
  BEZ235 (NVP-BEZ235) is a dual ATP-competitive PI3K and mTOR inhibitor. Inhibits ATR whileshown to be a poor inhibitor to Akt and PDK1.
  Patients will take the BEZ235 (capsules) orally with food. The dose should be taken every 3 weeks.
  Ipatasertib (GDC-0068) is a highly selective pan-Akt inhibitor targeting Akt1/2/3 .
  Patients will take the Ipatasertib (capsules) orally with food. The dose should be taken every 3 weeks.
  The suggested dosage of inhibitors of the PI3K/Akt pathway orally as a single dose in capsule and Packed in plastic boxes, so that preparations can be taken at home
  Interventions: Biological: Suppressor of the PI3K/Akt pathways

INTERVENTIONS:
Drug: MK - 3475 — Administered Intravenously
  Other Names: Pembrolizumab; Keytruda
  Arms: MK-3475
Biological: Suppressor of the PI3K/Akt pathways — Capsules orally with food
  Other Names: Pictilisib; GDC-0941; BEZ235; NVP-BEZ235; Ipatasertib; GDC-0068
  Arms: Suppressor of the PI3K/Akt pathways

SUMMARY:
It is known that after application of MK-3475 activated PD -1 negatively regulates the activation of T cells through suppression of the path of PI3K / Akt.

This study will identify the effectiveness of oral inhibitors of PI3K / Akt pathway in comparison with MK-3475 (pembrolizumab).

DETAILED DESCRIPTION:
A humanized monoclonal IgG4 antibody directed against human cell surface receptor PD-1 (programmed death-1 or programmed cell death-1) with potential immunopotentiating activity. Upon administration, pembrolizumab binds to PD-1, an inhibitory signaling receptor expressed on the surface of activated T cells, and blocks the binding to and activation of PD-1 by its ligands, which results in the activation of T-cell-mediated immune responses against tumor cells. The ligands for PD-1 include PD-L1, which is expressed on antigen presenting cells (APCs) and overexpressed on certain cancer cells, and PD-L2, which is primarily expressed on APCs. Activated PD-1 negatively regulates T-cell activation through the suppression of the PI3K/Akt pathway.

This study will identify the effectiveness of oral inhibitors of PI3K / Akt pathway in comparison with MK-3475 (pembrolizumab).

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed World Health Organization Grade IV malignant glioma (glioblastoma or gliosarcoma). Participants will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of glioblastoma or variants is made.
* Previous first line therapy with at least radiotherapy and temozolomide
* Be at first or second relapse.
* Participants must have shown unequivocal evidence for tumor progression by MRI or CT scan.
* CT or MRI within 14 days prior to start of study drug.
* An interval of at least 4 weeks (to start of study agent) between prior surgical resection or one week for stereotactic biopsy.
* An interval of at least 12 weeks from the completion of radiation therapy to start of study drug unless there is a new area of enhancement consistent with recurrent tumor outside the radiation field or there is unequivocal histologic confirmation of tumor progression
* Participants must have recovered to grade 0 or 1 or pre-treatment baseline from clinically significant toxic effects of prior therapy (including but not limited to exceptions of alopecia, laboratory values listed per inclusion criteria, and lymphopenia which is common after therapy with temozolomide).
* From the projected start of scheduled study treatment, the following time periods must have elapsed: 5 half-lives from any investigational agent, 4 weeks from cytotoxic therapy (except 23 days for temozolomide and 6 weeks from nitrosoureas), 6 weeks from antibodies, or 4 weeks (or 5 half-lives, whichever is shorter) from other anti-tumor therapies.
* Payment of charitable contributions may be required

Exclusion Criteria:

* Current or planned participation in a study of an investigational agent or using an investigational device.
* Has a diagnosis of immunodeficiency.
* Has tumor primarily localized to the brainstem or spinal cord.
* Has presence of diffuse leptomeningeal disease or extracranial disease.
* Has received systemic immunosuppressive treatments within 6 months of start of study drug
* Requires treatment with high dose systemic corticosteroids defined as dexamethasone > 4 mg/day or bioequivalent for at least 3 consecutive days within 2 weeks of start of study drug.
* Has received prior interstitial brachytherapy, implanted chemotherapy, stereotactic radiosurgery or therapeutics delivered by local injection or convection enhanced delivery.
* Requires therapeutic anticoagulation with warfarin at baseline; patients must be off warfarin or warfarin-derivative anti-coagulants for at least 7 days prior to starting study drug; however, therapeutic or prophylactic therapy with low-molecular weight heparin is allowed.
* Has history of known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhage within 12 months of start of study drug
* Has evidence of intratumoral or peritumoral hemorrhage on baseline MRI scan other than those that are grade ≤ 1 and either post-operative or stable on at least 2 consecutive MRI scans.
* Has gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE Grade > 3 within 6 months of start of study drug.
* Has a known additional malignancy that is progressing or requires active treatment within 3 years of start of study drug. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial
* Has a known history of HIV
* Has known active Hepatitis B or Hepatitis C
* Has received a live vaccine within 30 days prior to the first dose of study drug.
* Has a known hypersensitivity to any of the study therapy products.
* Has received anti-angiogenic or anti-VEGF targeted agents (e.g. bevacizumab, cediranib, aflibercept, vandetanib, XL-184, sunitinib, etc)
* Has a history of non-healing wounds or ulcers, or bone refractures within 3 months of fracture
* Has a history of arterial thromboembolism within 12 months of start of study drug.
* Has inadequately controlled hypertension
* Has a history of hypertensive crisis or hypertensive encephalopathy
* Has had clinically significant cardiovascular disease within 12 months of start of study drug
* Has a history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to start of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-01 (Actual); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Time Frame: 12 months
  To evaluate the anti-tumor activity of pembrolizumab among subjects with recurrent glioblastoma when treated with pembrolizumab (Cohort A), and when treated with inhibitors PI3K/Akt pathways monotherapy (Cohort B) as assessed by the 12-month progression-free survival (PFS-12) rate.

SECONDARY OUTCOMES:
Safety and tolerability of Pembrolizumab (Assessed by reported adverse events using CTCAE version 4.0) | Time Frame: 12 months
  Assesed by reported adverse events using CTCAE version 4.0. Progression Free Survival

OTHER OUTCOMES:
Safety and tolerability of inhibitors PI3K/Akt pathways as monotherapy (adverse events using CTCAE version 4.0) | Time Frame: 12 months
  Assesed by reported adverse events using CTCAE version 4.0. Progression Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Jann Lee, PhD, Principal Investigator — MRC Clinical Trials Unit
Locations (13):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - M D Anderson Cancer Center, Houston, Texas
- UCL- Cliniques Universitaires Saint Luc, Brussels, Belgium
- St Johannes Hospital, Duisburg, Germany
- Italy (2):
  - Spedali Civili di Brescia, Brescia
  - IRCCS San Raffaele, Milan
- Lower-Silesian Oncology Centre, Wroclaw, Lower Silesian Voivodeship, Poland
- Pavlov State Medical University, Saint Petersburg, Russia
- Hospital Universitario Germans Trias I Pujol, Barcelona, Spain
- Universitätsklinik für Frauenheilkunde, Bern, Switzerland
- Ukraine (2):
  - Regional Cancer Center, Dnipro
  - National Institute of Cancer, Kiev
- Royal Victoria Hospital, Belfast, Ulster, United Kingdom